CLINICAL TRIAL: NCT03774927
Title: A Randomized, Double-blind Sham-controlled Trial of High Frequency rTMS for Cognitive Impairments in Chronic Schizophrenia Patients
Brief Title: High Frequency rTMS Treatment for Cognitive Impairments in Chronic Schizophrenia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, Professor, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CASPsy1
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; rTMS
MeSH Terms: conditions — Schizophrenia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10 Hz treatment group (Experimental): In active rTMS, 10 Hz stimulations over left DLPFC occurred at a power of 110% of MT for 27-s intervals with 20s inter-train interval. 20 minutes were administered each day (Monday-Friday) for 8 consecutive weeks.
  Interventions: Device: 10 Hz treatment group
- 20 Hz treatment group (Experimental): In active rTMS, 20 Hz stimulations over left DLPFC occurred at a power of 110% of MT for 20 intervals with 28s inter-train interval. 20 minutes were administered each day (Monday-Friday) for 8 consecutive weeks.
  Interventions: Device: 20 Hz treatment group
- Control Group (Sham Comparator): In sham rTMS, all procedures were identical to 10Hz group except they were the non-magnetized steel cylinders, instead of cylindrical magnets, that were rotated.
  Interventions: Device: Control Group

INTERVENTIONS:
Device: 10 Hz treatment group — 10 Hz stimulations over left DLPFC occurred at a power of 110% of MT for 27-s intervals with 20s inter-train interval. 20 minutes were administered each day (Monday-Friday) for 8 consecutive weeks.
  Arms: 10 Hz treatment group
Device: 20 Hz treatment group — 20 Hz stimulations over left DLPFC occurred at a power of 110% of MT for 20 intervals with 28s inter-train interval. 20 minutes were administered each day (Monday-Friday) for 8 consecutive weeks.
  Arms: 20 Hz treatment group
Device: Control Group — all procedures were identical to 10Hz group except they were the non-magnetized steel cylinders, instead of cylindrical magnets, that were rotated.
  Arms: Control Group

SUMMARY:
A randomized, double-blind sham-controlled trial of high frequency rTMS treatment for cognitive impairments in 120 chronic schizophrenia patients

DETAILED DESCRIPTION:
OBJECTIVE: This study aimed to evaluate the efficacy of high-frequency repetitive transcranial magnetic stimulation (rTMS) over left dorsolateral prefrontal cortex in the treatment of cognitive impairments in 120 chronic patients with schizophrenia.

METHODS:

1. Clinical Trial: The study consists of 8 weeks of treatment.
2. Assessment Procedures:

2.1 Primary Outcome Variable-Psychopathology: The psychopathology of patients was assessed by three clinical trained staff, who were blind to treatment protocols, using the Positive and Negative Syndrome Scale (PANSS). Patients are interviewed at screening, at at baseline, 2 weeks, 4 weeks, 6 weeks and 8 weeks.

2.2 Cognitive tests: RBANS was used to assess the cognitive function by three psychologists, which is comprised of a total score and 5 age-adjusted index scores for attention, language, delayed and immediate memory and visuospatial/construction. A translated and adapted Chinese version of RBANS has been evaluated for the test-retest reliability and clinical validity between schizophrenia patients and control subjects. Cognitive performance was measured at baseline and at 8-weeks.

2.3 Side Effects: TESS was used to assess the side effect at baseline and every 2 weeks.

2.5 Weight gain measurement: weight gain every week

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizopherenia by two senior psychiatrists
* Male
* Right-handed
* Between 18 and 60 years and Han Chinese
* Duration of symptoms at least 60 months
* Received stable doses of antipsychotic drugs at least 12 months
* With unresolved negative symptoms (Negative scale of PANSS ≥20 and positive scale of PANSS < 24)

Exclusion Criteria:

* A DSM-IV Axis I diagnosis other than schizophrenia
* Documented disease of physical diseases including, but not limited to seizure, epilepsy, aneurysm brain tumor, and stroke, dementia, parkinson's disease, Huntington's disease, multiple sclerosis
* Acute, unstable and/or significant and untreated medical illness (e.g., infection, unstable diabetes, uncontrolled hypertension)
* Severe headache for unknown reasons and cardiovascular diseases, intra-cranial metals, pacemakers, severe and those receiving electroconvulsive therapy in the past 3 months
* Past history of autoimmune and allergies, hypertension, lung disease, diabetes or cerebrovascular disease), past history of neurological illness (head trauma with loss of consciousness for more than 5 minutes) or family history of epilepsy increasing the risk of seizures
* Education level less than 5 years by subject report,
* Receiving or planning to start the psychotherapy during the rTMS treatment or past received psychotherapy 6 months before the current study
* Subjects who suffered from alcohol or illegal drug abuse/dependence

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Repeatable Battery for the Assessment of Neuropsychological Status for cognition | 8 weeks
  cognitive performance
Positive and Negative Syndrome Scale for clinical symptoms | 8 weeks
  clinical symptoms

SECONDARY OUTCOMES:
Treatment Emergent Symptoms Scale for side effects | 8 weeks
  Side effect

CONTACTS AND LOCATIONS:
Overall Officials: Hengyong Guan, Doctor, Principal Investigator — Hebei Province Veteran Psychiatric Hospital

IPD SHARING:
Plan to Share IPD: No
Data with be available on request

REFERENCES:
- [Background] Dlabac-de Lange JJ, Liemburg EJ, Bais L, Renken RJ, Knegtering H, Aleman A. Effect of rTMS on brain activation in schizophrenia with negative symptoms: A proof-of-principle study. Schizophr Res. 2015 Oct;168(1-2):475-82. doi: 10.1016/j.schres.2015.06.018. Epub 2015 Jul 14. PMID 26187147
- [Result] Mogg A, Purvis R, Eranti S, Contell F, Taylor JP, Nicholson T, Brown RG, McLoughlin DM. Repetitive transcranial magnetic stimulation for negative symptoms of schizophrenia: a randomized controlled pilot study. Schizophr Res. 2007 Jul;93(1-3):221-8. doi: 10.1016/j.schres.2007.03.016. Epub 2007 May 2. PMID 17478080
- [Result] Wobrock T, Guse B, Cordes J, Wolwer W, Winterer G, Gaebel W, Langguth B, Landgrebe M, Eichhammer P, Frank E, Hajak G, Ohmann C, Verde PE, Rietschel M, Ahmed R, Honer WG, Malchow B, Schneider-Axmann T, Falkai P, Hasan A. Left prefrontal high-frequency repetitive transcranial magnetic stimulation for the treatment of schizophrenia with predominant negative symptoms: a sham-controlled, randomized multicenter trial. Biol Psychiatry. 2015 Jun 1;77(11):979-88. doi: 10.1016/j.biopsych.2014.10.009. Epub 2014 Oct 23. PMID 25582269
- [Derived] Zhu C, Yao J, Guan H, Wu F, Xiu M. Moderating role of familial relationships in the efficacy of rTMS intervention on cognitive function in patients with schizophrenia. BMC Psychiatry. 2025 Oct 21;25(1):1010. doi: 10.1186/s12888-025-07251-y. PMID 41121094
- [Derived] Su X, Zhao L, Shang Y, Chen Y, Liu X, Wang X, Xiu M, Yu H, Liu L. Repetitive transcranial magnetic stimulation for psychiatric symptoms in long-term hospitalized veterans with schizophrenia: A randomized double-blind controlled trial. Front Psychiatry. 2022 Sep 23;13:873057. doi: 10.3389/fpsyt.2022.873057. eCollection 2022. PMID 36213928
- [Derived] Xiu MH, Guan HY, Zhao JM, Wang KQ, Pan YF, Su XR, Wang YH, Guo JM, Jiang L, Liu HY, Sun SG, Wu HR, Geng HS, Liu XW, Yu HJ, Wei BC, Li XP, Trinh T, Tan SP, Zhang XY. Cognitive Enhancing Effect of High-Frequency Neuronavigated rTMS in Chronic Schizophrenia Patients With Predominant Negative Symptoms: A Double-Blind Controlled 32-Week Follow-up Study. Schizophr Bull. 2020 Sep 21;46(5):1219-1230. doi: 10.1093/schbul/sbaa035. PMID 32185388